CLINICAL TRIAL: NCT05200169
Title: An Open-Label, Non-Randomised, Single-Dose, Single-Period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of 14C-AB1010 in Healthy Male Subjects
Brief Title: Mass Balance Recovery, Metabolite Profile and Metabolite Identification of 14C-AB1010 in Healthy Male Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB17001; 2017-001948-34 (EudraCT Number)
Record Dates: First submitted 2021-12-27; First posted 2022-01-20 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: An open label, non-randomized, single-dose, single-period study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 14C-AB1010 (Experimental): Oral solution of 14C radiolabelled AB1010 (200 mg per subject)
  Interventions: Drug: 14C-AB1010

INTERVENTIONS:
Drug: 14C-AB1010 — Oral solution of 14C radiolabelled AB1010 (200 mg per subject)
  Other Names: radiolabelled masitinib

SUMMARY:
To assess the mass balance recovery after a single oral dose of 14C-AB1010

DETAILED DESCRIPTION:
The objective is to characterize the distribution, metabolism and elimination of AB1010 in humans through the sampling of blood, urine, and faeces. This is accomplished through the administration of 14C-AB1010 oral solution with a therapeutic relevant dose of AB1010 as a single oral dose. There was no control group and no blinding as the objective was to assess the mass balance of masitinib after a single oral intake. There was only one group of healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria Included:

* Healthy Male as determined by a physician, based on a medical evaluation including medical history, physical examination, clinical laboratory tests and 12-lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the Sponsor Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male between 18 and 65 years old inclusive, at the time of signing the informed consent.
* Body mass index of 18.0 to 32.0 kg/m2, inclusive at screening
* Body weight between 60 and 90 kg
* Normal blood pressure and heart rate or, if abnormal, considered not clinically significant by the principal Investigator or sub-investigator.
* Neutrophils count should be within normal range or deemed as not clinically significant by the PI
* Must have regular bowel movements (ie, average stool production of ≥1 and ≤3 stools per day)

Exclusion Criteria Included:

* Any clinically significant cardio vascular diseases such as but not limited to the common reported below:

  * History or presence or suspect of Acute Coronary Syndrome, Myocardial Infarction, Coronary Artery bypass graft surgery or stent procedure;
  * History or presence or suspect of Angina Pectoris;
  * History or presence or suspect, heart failure;
  * Abnormal vital signs
  * Clinically significant abnormal Blood Pressure according to investigator's opinion
  * Abnormal resting ECG according investigator's opinion.
* Clinically significant, abnormal medical history, physical findings, ECG, or laboratory values at the screening visit that could interfere with the objectives of the study or the safety of the volunteer.
* A history of clinically significant acute illness (resolved within 4 weeks of screening), or history of significant cardiac arrhythmias or unexplained syncope or presence of cardiovascular, gastrointestinal, renal, hepatic, neurologic, haematologic, endocrine, oncologic, pulmonary, immunologic, dermatologic or psychiatric disease or any other condition which, in the opinion of the Principal Investigator (PI), would jeopardize the safety of the subject or impact the validity of the study results.
* Subject has an uncontrolled intercurrent illness (i.e., active infection) or fever (oral temperature > 38 degrees Celsius) at screening.
* Clinically significant history of or current seizure disorder or history of syncope, unexplained loss of consciousness or clinically significant history of Central Nervous System (CNS) disorders
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Radioactivity recovery | 168 hours post-dose
  Cumulative Amount of Total Radioactivity Excreted in Urine. No statistical analyses have been specified for this primary end point. It is expected there is at least one statistical analysis for each primary end point. No formal statistical analysis were performed for this study due to the small number of subjects, for which statistical inference is not meaningful.

CONTACTS AND LOCATIONS:
Overall Officials: Nand Singh, MD, Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Masitinib is under clinical investigation and has not yet been approved in any sought-after indication by any health authority worldwide. As such, there is no plan for data-sharing at this point in time.